CLINICAL TRIAL: NCT06256081
Title: Testing the Hear Glue Ear Software Application on Patients With Glue Ear
Brief Title: Testing a New App for Children With Glue Ear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Tamsin Brown (Other)
Responsible Party: Sponsor-Investigator, Dr. Tamsin Brown, Principal investigator, Cambridgeshire Community Services NHS Trust
Organization: Cambridgeshire Community Services NHS Trust (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 262154
Record Dates: First submitted 2019-02-25; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Hearing Loss, Conductive
Keywords: glue ear
MeSH Terms: conditions — Hearing Loss, Conductive; Otitis Media with Effusion

STUDY DESIGN:
Intervention Model Description: Teal of an app
Masking Description: Single arm study of children trialling an app
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children with hearing loss secondary to glue ear (Active Comparator): Children accessing the community audiology NHS services due to concerns about hearing loss who have a diagnosis of glue ear (also known as otitis media with effusion, OME)
  Interventions: Device: Hear Glue ear application
- Children with normal hearing (Sham Comparator): Children accessing the community audiology NHS services due to concerns about hearing loss who do not have a diagnosis of glue ear (also known as otitis media with effusion, OME) and are confirmed as having normal hearing.
  Interventions: Device: Hear Glue ear application

INTERVENTIONS:
Device: Hear Glue ear application — Hear Glue ear is an application used on phones, ipads, tablets or computers which provides free information, songs, audiobooks, games and a home hearing screening game.
  Other Names: headphones used with the hearing screening game on the application

SUMMARY:
To assess whether children with glue ear ( and some normal hearing controls) and their families find the Hear Glue Ear application acceptable and easy to use. Whether the hearing screening section on the app is comparable to the hearing test data obtained from formal audiology hearing tests.

DETAILED DESCRIPTION:
The Hear Glue Ear application aims to provide up-to-date information for families as well as audiobooks, songs and games for children with hearing loss secondary to glue ear, to be able to aid with their developmental skills (particularly speech, language, auditory processing, auditory memory and listening skills) during the period of time when they have glue ear.

Outcome measures include acceptability of the application by the family (provided by questionnaires to the child and an adult parent/ carer), usability of the app (a member of the research team will observe the child using the app and how much difficulty they have such as how many times the researcher has to help/ intervene) and comparison of the hearing screen on the app with formal audiology hearing test result.

ELIGIBILITY:
Inclusion Criteria:

* aged 2-8 years old
* had a formal hearing test at Cambridge audiology clinic and has a diagnosis of gluem ear worse than 25dB at more than 1 frequency or nornmal hearing diagnosed where 20dB or better is recorded at 0.5, 1, 2, 4 KHz

Exclusion Criteria:

* permanent hearing loss
* English not a dominant language (since the app is written in English)

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
acceptability of the Hear Glue Ear application to children with glue ear and their families | Observing the child looking at the app for he first time and following up with the family after 1 week from baseline regarding whether they used it at home
  Questionnaire: Whether children like the Hear Glue ear app and find it useful

SECONDARY OUTCOMES:
does the hearing screen on the Hear Glue Ear application compare to hearing test results from formal audiology testing. | 1 hour maximum. one appointmnet where the researcher observes the child accessing the app
  Comparison between results: Children will have had a formal hearing test before they are invited into the study and theis will be compared to their results on the hearing screening game within the application.
Ease of use of the Hear Glue ear application | 1 hour. one appointmnet where the researcher observes the child accessing the app
  Questionnaire and Number of mistakes: Can children easily access the Hear Glue Ear application without help from an adult

CONTACTS AND LOCATIONS:
Overall Officials: Tamsin Holland Brown, MBBS, Principal Investigator — Cambridgeshire Community Services
Locations (1):
- Cambridgshire Community Services NHS Trust, Cambridge, Cambridgshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All patient data will only be held by the small research team gathering data for this project. Data will be held in line with GDPR and ethical approval.

REFERENCES:
- See also: Website used to give information about study outcomes to participants — http://www.hearglueear.Wordpress.com